CLINICAL TRIAL: NCT03209323
Title: Influence of Volatile Induction of General Anaesthesia With Sevoflurane Using Two Different Techniques and Intravenous Induction Using Propofol on the Epileptiform Electroencephalograph Patterns:
Brief Title: Epileptiform EEG Patterns During Induction of General Anaesthesia With Sevoflurane Compared to Those With Propofol
Acronym: EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Principal Investigator, Michał Stasiowski, Principal Investigator, Department of Anaesthesiology and Intensive Therapy, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SilesianMUKOAIIT6
Record Dates: First submitted 2017-07-02; First posted 2017-07-06 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: General Anaesthesia; Depth of Anaesthesia; Intraoperative Awareness; Seizures; Electroencephalography
Keywords: Epileptiform patterns; sevoflurane; propofol; bispectral index; state entropy; response entropy; A-line Auto Regressive Index; middle latency auditory evoked potentials
MeSH Terms: conditions — Intraoperative Awareness; Seizures | interventions — Electroencephalography; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant
Masking Description: The EEGs recorded before and during the general anaesthesia induction analysed offline by a neurophysiologist with an expertise in anaesthetic EEGs, the recording technique, and the anaesthetic agent used unaware of group allocation of the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sevoflurane - increasing concentrations (Experimental): The patient was breathing spontaneously via the face mask and the sevoflurane concentration in the inhaled gas was doubled every 10 breaths starting from 0.3 vol. % in a sequence 0.3-0.6-1.2-2.4-4.8-8 vol. % until a minimal alveolar concentration (MAC) of 2 was obtained in the exhalation gas. Electroencephalography (EEG), bispectral index (BIS), response and state entropy (RE and SE), middle latency auditory evoked potentials (MLAEP) were monitored.
  Interventions: Device: electroencephalography (EEG); Device: bispectral index (BIS); Device: response and state entropy (RE and SE); Device: middle latency auditory evoked potentials (MLAEP)
- sevoflurane - vital capacity (Experimental): The anaesthetic circuit was prefilled with 8% sevoflurane. The patients were asked to exhale to the residual volume. Then the patients were explained to perform a vital-capacity breath with a face mask applied tightly to their faces. Then the patients were encouraged to hold their breaths as long as possible. Thereafter, the patients were asked to breathe spontaneously. Electroencephalography (EEG), bispectral index (BIS), response and state entropy (RE and SE), middle latency auditory evoked potentials (MLAEP) were monitored.
  Interventions: Device: electroencephalography (EEG); Device: bispectral index (BIS); Device: response and state entropy (RE and SE); Device: middle latency auditory evoked potentials (MLAEP)
- propofol - intravenous induction (Experimental): the patients were preoxygenated with 100% oxygen following which propofol was intravenously administered at a single dose of 2.5 mg/kg of body weight, after which it was infused with an infusion speed of 4 mg/kg body weight/h. Electroencephalography (EEG), bispectral index (BIS), response and state entropy (RE and SE), middle latency auditory evoked potentials (MLAEP) were monitored.
  Interventions: Device: electroencephalography (EEG); Device: bispectral index (BIS); Device: response and state entropy (RE and SE)

INTERVENTIONS:
Device: electroencephalography (EEG) — Four EEG channels were recorded using electrode positions as defined in the International 10-20 System with Ag/AgCl2 cup electrodes (Spes Medica) attached to the scalp with EC2 Electrode Cream (Grass Technologies). The impedance was set below 1 k, and the electrodes were attached to module S/5 E-EEG of the anaesthetic monitor S/5 (GE Healthcare).
Device: bispectral index (BIS) — The BIS score was derived from a sensor (Aspect Medical Systems) positioned diagonally on the patients' foreheads according to producer's instructions.
Device: response and state entropy (RE and SE) — The respone and state entropy (RE and SE) score was derived from a sensor (Aspect Medical Systems) positioned diagonally on the patients' foreheads according to producer's instructions.
Device: middle latency auditory evoked potentials (MLAEP) — value of A-line Auto Regressive Index (AAI) derived from middle latency auditory evoked potentials (MLAEP) (A-line Monitor, Danmeter A/S, Odense, Denmark) was observed which measures the central nervous system responsiveness to a specific auditory stimulus
  Arms: sevoflurane - increasing concentrations; sevoflurane - vital capacity

SUMMARY:
The aim of the study was to assess the influence of volatile induction of general anaesthesia with sevoflurane using two different techniques and intravenous anaesthesia with propofol on the possible presence of epileptiform electroencephalograph patterns during the induction of general anaesthesia. We aimed to verify whether presence of epileptiform patterns (EPs) defined as polispikes (PS), rhytmic polispikes (RPS), periodic epileptiform discharges (PED) on Electroencephalographs (EEGs) influence the behaviour of values of the Bispectral Index (BIS), State (SE) and Response (RE), A-line Auto Regressive Index (AAI) derived from middle latency auditory evoked potentials (MLAEP) during the induction of general anaesthesia using abovementioned techniques and such variations may be useful in detection of presence of EPs.

DETAILED DESCRIPTION:
Both sevoflurane and propofol are considered safe and potent anaesthetics and are used for induction or coinduction of general anaesthesia. During all stages of general anaesthesia, both agents may induce seizure-like movements or seizures (clinically manifested events and confirming electroencephalographic pattern) accompanied by haemodynamic instability. Their proconvulsant activity should be verified and assessed.

The aim of the additional analysis was to identify whether observance of the variations of values displayed on different depth of anaesthesia monitors (DOA monitors) reliably reflect the actual depth of general anaesthesia during presence of epileptiform patterns (EPs) in EEGs during VIGA with sevoflurane using two different techniques and intravenous induction of general anaesthesia with single dose of propofol.

We performed standard 30-minute initial EEG recordings for all patients participating in the study to exclude any pre-existing epileptic EEG patterns. We took the initial EEG recordings in a dark quiet room for 5 minutes as a baseline, followed by three eye opening and closing sequences of 10 seconds each and photostimulation lasting 10 minutes (flash stimuli at frequencies of 3/6/9/12 Hz- alpha; 15/18/21/24 Hz- beta). Then we obtained another baseline reading and we asked the patients to achieve a state of hyperventilation by taking 20 forceful breathes per minute for five minutes. Finally, we obtained another baseline reading.

Throughout the induction of anaesthesia and the surgery, standard monitoring procedures were utilised to pay close attention to the vital parameters such as non-invasive arterial pressure (BP), heart rate (HR), standard electrocardiography (ECG) II, arterial oxygen saturation (SaO2), fraction of inspired oxygen in the gas mixture (FiO2), facial electromyography (fEMG), fraction of inspired sevoflurane (FiAA), fraction of expired sevoflurane (FeAA), exhaled carbon dioxide concentration (etCO2), minimal alveolar concentration of sevoflurane (MAC).

ELIGIBILITY:
Inclusion Criteria:

* an American Society of Anaesthesiologists (ASA) score I-II
* written informed consent to undergo general anaesthesia

Exclusion Criteria:

- history of epilepsy, medical treatment that might interfere with the EEG (e.g., tranquilizers, antiepileptic drugs), pregnancy, drug or alcohol abuse, history of neurological disease or a neurosurgical operation that would impair EEG or BIS monitoring, history of pulmonary disease, or the presence of signs predicting difficult mask ventilation or intubation. any pre-existing epileptic EEG patterns in standard 30-minute initial EEG recordings performed in all the patients participating in the study.

Ages: 18 Years to 70 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2008-12-13 (Actual); Study Completion 2008-12-13 (Actual)

PRIMARY OUTCOMES:
presence of epileptiform patterns in patients EEGs | intraoperative
  the main objective is to measure the influence of volatile induction of general anaesthesia with sevoflurane using two different techniques and intravenous anaesthesia with propofol on the presence of epileptiform electroencephalograph patterns during the induction of general anaesthesia.

SECONDARY OUTCOMES:
observance of BIS score behaviour during presence of epileptiform patterns in patients EEGs | intraoperative
  the objective is to measure the BIS index variations during presence of EPs in patients' EEGs during volatile induction of general anaesthesia (VIGA) with sevoflurane using two different anaesthetic regimens compared to intravenous induction of general anaesthesia using single dose of propofol.
observance of values of state and response entropy behaviour during presence of epileptiform patterns in patients | intraoperative
  the objective is to measure values of state and response entropy index variations during presence of EPs in patients' EEGs during volatile induction of general anaesthesia (VIGA) with sevoflurane using two different anaesthetic regimens compared to intravenous induction of general anaesthesia using single dose of propofol.
observance of values of middle latency auditory evoked potentials behaviour during presence of epileptiform patterns in patients | intraoperative
  the objective is to measure values of middle latency auditory evoked potentials during presence of EPs in patients' EEGs during volatile induction of general anaesthesia (VIGA) with sevoflurane using two different anaesthetic regimens compared to intravenous induction of general anaesthesia using single dose of propofol.

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Jałowiecki, Principal Investigator — Silesian University of Medicine
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
articles in Clinical Monitoring and Computing in 2017, case reports

REFERENCES:
- [Background] Viertio-Oja H, Maja V, Sarkela M, Talja P, Tenkanen N, Tolvanen-Laakso H, Paloheimo M, Vakkuri A, Yli-Hankala A, Merilainen P. Description of the Entropy algorithm as applied in the Datex-Ohmeda S/5 Entropy Module. Acta Anaesthesiol Scand. 2004 Feb;48(2):154-61. doi: 10.1111/j.0001-5172.2004.00322.x. No abstract available. PMID 14995936
- [Result] Chinzei M, Sawamura S, Hayashida M, Kitamura T, Tamai H, Hanaoka K. Change in bispectral index during epileptiform electrical activity under sevoflurane anesthesia in a patient with epilepsy. Anesth Analg. 2004 Jun;98(6):1734-1736. doi: 10.1213/01.ANE.0000117282.72866.26. PMID 15155337
- [Result] Sarkela MO, Ermes MJ, van Gils MJ, Yli-Hankala AM, Jantti VH, Vakkuri AP. Quantification of epileptiform electroencephalographic activity during sevoflurane mask induction. Anesthesiology. 2007 Dec;107(6):928-38. doi: 10.1097/01.anes.0000291444.68894.ee. PMID 18043061
- [Result] Gibert S, Sabourdin N, Louvet N, Moutard ML, Piat V, Guye ML, Rigouzzo A, Constant I. Epileptogenic effect of sevoflurane: determination of the minimal alveolar concentration of sevoflurane associated with major epileptoid signs in children. Anesthesiology. 2012 Dec;117(6):1253-61. doi: 10.1097/ALN.0b013e318273e272. PMID 23103557
- [Result] Kreuzer I, Osthaus WA, Schultz A, Schultz B. Influence of the sevoflurane concentration on the occurrence of epileptiform EEG patterns. PLoS One. 2014 Feb 26;9(2):e89191. doi: 10.1371/journal.pone.0089191. eCollection 2014. PMID 24586585
- [Result] Jaaskelainen SK, Kaisti K, Suni L, Hinkka S, Scheinin H. Sevoflurane is epileptogenic in healthy subjects at surgical levels of anesthesia. Neurology. 2003 Oct 28;61(8):1073-8. doi: 10.1212/01.wnl.0000090565.15739.8d. PMID 14581667
- [Result] Pilge S, Jordan D, Kochs EF, Schneider G. Sevoflurane-induced epileptiform electroencephalographic activity and generalized tonic-clonic seizures in a volunteer study. Anesthesiology. 2013 Aug;119(2):447. doi: 10.1097/ALN.0b013e31827335b9. No abstract available. PMID 23221897
- [Result] Kaisti KK, Jaaskelainen SK, Rinne JO, Metsahonkala L, Scheinin H. Epileptiform discharges during 2 MAC sevoflurane anesthesia in two healthy volunteers. Anesthesiology. 1999 Dec;91(6):1952-5. doi: 10.1097/00000542-199912000-00052. No abstract available. PMID 10598642
- [Result] Vakkuri A, Jantti V, Sarkela M, Lindgren L, Korttila K, Yli-Hankala A. Epileptiform EEG during sevoflurane mask induction: effect of delaying the onset of hyperventilation. Acta Anaesthesiol Scand. 2000 Jul;44(6):713-9. doi: 10.1034/j.1399-6576.2000.440609.x. PMID 10903015
- [Result] Julliac B, Guehl D, Chopin F, Arne P, Burbaud P, Sztark F, Cros AM. Risk factors for the occurrence of electroencephalogram abnormalities during induction of anesthesia with sevoflurane in nonepileptic patients. Anesthesiology. 2007 Feb;106(2):243-51. doi: 10.1097/00000542-200702000-00011. PMID 17264717
- [Result] Ben-Menachem E, Zalcberg D. Depth of anesthesia monitoring: a survey of attitudes and usage patterns among Australian anesthesiologists. Anesth Analg. 2014 Nov;119(5):1180-5. doi: 10.1213/ANE.0000000000000344. PMID 25006849
- [Result] Vakkuri A, Yli-Hankala A, Sarkela M, Lindgren L, Mennander S, Korttila K, Saarnivaara L, Jantti V. Sevoflurane mask induction of anaesthesia is associated with epileptiform EEG in children. Acta Anaesthesiol Scand. 2001 Aug;45(7):805-11. doi: 10.1034/j.1399-6576.2001.045007805.x. PMID 11472278
- [Result] Yli-Hankala A, Vakkuri A, Sarkela M, Lindgren L, Korttila K, Jantti V. Epileptiform electroencephalogram during mask induction of anesthesia with sevoflurane. Anesthesiology. 1999 Dec;91(6):1596-603. doi: 10.1097/00000542-199912000-00009. PMID 10598599
- [Result] Aho AJ, Yli-Hankala A, Lyytikainen LP, Jantti V. Facial muscle activity, Response Entropy, and State Entropy indices during noxious stimuli in propofol-nitrous oxide or propofol-nitrous oxide-remifentanil anaesthesia without neuromuscular block. Br J Anaesth. 2009 Feb;102(2):227-33. doi: 10.1093/bja/aen356. Epub 2008 Dec 25. PMID 19112059
- [Result] Jensen EW, Lindholm P, Henneberg SW. Autoregressive modeling with exogenous input of middle-latency auditory-evoked potentials to measure rapid changes in depth of anesthesia. Methods Inf Med. 1996 Sep;35(3):256-60. PMID 8952311
- [Result] Newton DE, Thornton C, Konieczko KM, Jordan C, Webster NR, Luff NP, Frith CD, Dore CJ. Auditory evoked response and awareness: a study in volunteers at sub-MAC concentrations of isoflurane. Br J Anaesth. 1992 Aug;69(2):122-9. doi: 10.1093/bja/69.2.122. PMID 1389813
- [Result] Gajraj RJ, Doi M, Mantzaridis H, Kenny GN. Comparison of bispectral EEG analysis and auditory evoked potentials for monitoring depth of anaesthesia during propofol anaesthesia. Br J Anaesth. 1999 May;82(5):672-8. doi: 10.1093/bja/82.5.672. PMID 10536541
- [Result] Schraag S, Bothner U, Gajraj R, Kenny GN, Georgieff M. The performance of electroencephalogram bispectral index and auditory evoked potential index to predict loss of consciousness during propofol infusion. Anesth Analg. 1999 Nov;89(5):1311-5. PMID 10553858
- [Result] Pilge S, Kreuzer M, Karatchiviev V, Kochs EF, Malcharek M, Schneider G. Differences between state entropy and bispectral index during analysis of identical electroencephalogram signals: a comparison with two randomised anaesthetic techniques. Eur J Anaesthesiol. 2015 May;32(5):354-65. doi: 10.1097/EJA.0000000000000189. PMID 25564779